CLINICAL TRIAL: NCT05498129
Title: School Feeding to Improve Cognitive Performance in Disadvantaged Children: A Randomized Controlled Trial in in Northwest Pakistan
Brief Title: School Feeding to Improve Cognitive Performance in Disadvantaged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: Khyber Medical University (Unknown)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: School Feeding
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No school meal (Active Comparator)
  Interventions: Other: No school meal
- School meal (Experimental)
  Interventions: Other: School meal
- School meal plus micronutrient powder (Experimental)
  Interventions: Other: School meal plus micronutrient powder

INTERVENTIONS:
Other: School meal — School lunch was comprised of rice, ghee and beef
  Arms: School meal
Other: School meal plus micronutrient powder — School lunch plus micronutrient powder
  Arms: School meal plus micronutrient powder
Other: No school meal — No school meal
  Arms: No school meal

SUMMARY:
This trial investigated the impact of providing a regular meal with and without additional multiple micronutrients for children in Northwest Pakistan on their performance at school, in comparison to a local government school that served as a control i.e. no school meal.

ELIGIBILITY:
Inclusion Criteria:

* Prep or class 1
* Male/ female

Exclusion Criteria:

* Any contraindicating condition

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Ravens Colour Matrices test for assessment of Cognitive function | Baseline
  Raven's Coloured Progressive Matrices. Raven's Coloured Progressive Matrices (RCPM) (20)is a widely used nonverbal intelligence test for children between the ages of 5 and 11 years. The test comprises 36-items in the form of three sets of 12 items, that increase in difficulty
Ravens Colour Matrices test for assessment of Cognitive function | 6-months
  Raven's Coloured Progressive Matrices. Raven's Coloured Progressive Matrices (RCPM) (20)is a widely used nonverbal intelligence test for children between the ages of 5 and 11 years. The test comprises 36-items in the form of three sets of 12 items, that increase in difficulty
Ravens Colour Matrices test for assessment of Cognitive function | 12-months
  Raven's Coloured Progressive Matrices. Raven's Coloured Progressive Matrices (RCPM) (20)is a widely used nonverbal intelligence test for children between the ages of 5 and 11 years. The test comprises 36-items in the form of three sets of 12 items, that increase in difficulty

SECONDARY OUTCOMES:
Height | Baseline
  Stature measured via a stadiometer
Mass | Baseline
  Body mass using a weighing scale
Mid upper arm circumference | Baseline
  Arm circumference
Height for age | Baseline
  Height for age calculated using the WHO calculator based on the 2006 WHO Child Growth Standards.
Weight for age | Baseline
  Weight for age calculated using the WHO calculator based on the 2006 WHO Child Growth Standards.
Haemoglobin | 6-months
  Haemoglobin measured by finger prick blood samples
Haemoglobin | 12-months
  Haemoglobin measured by finger prick blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Jonathan Sinclair, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No